CLINICAL TRIAL: NCT00329446
Title: A Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, Active-Controlled Study of the Efficacy and Safety of Sustained-Release Quetiapine Fumarate (SEROQUEL®) Compared With Placebo in the Treatment of Generalized Anxiety Disorder
Brief Title: Safety & Efficacy Study of Quetiapine Fumarate (SEROQUEL®) vs. Placebo & Active Control in Generalized Anxiety Disorder
Acronym: GOLD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1448C00010; GOLD
Record Dates: First submitted 2006-05-22; First posted 2006-05-24 (Estimated); Last update posted 2009-03-25 (Estimated); Status verified 2009-03

CONDITIONS: Generalized Anxiety Disorder
Keywords: GAD; anxiety
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety Disorders | interventions — Quetiapine Fumarate

INTERVENTIONS:
Drug: Quetiapine Fumarate
Drug: Escitalopram oxylate

SUMMARY:
The purpose of this study is to demonstrate that quetiapine SR (SEROQUEL®) is efficacious and safe in the acute treatment of patients with Generalized Anxiety Disorder.

PLEASE NOTE: Seroquel SR and Seroquel XR refer to the same formulation. The SR designation was changed to XR after consultation with FDA.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a documented clinical diagnosis of Generalized Anxiety Disorder.
* Be able to understand and comply with the requirements of the study.
* Able to understand and provide written informed consent

Exclusion Criteria:

* Patients (female) must not be pregnant or lactating
* Current or past diagnosis of stroke or transient ischemic attack (TIA).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2006-04; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Change from randomization in the HAM-A total score at Day 57

SECONDARY OUTCOMES:
Change from randomization in CGI-S score at Day 57

CONTACTS AND LOCATIONS:
Overall Officials: Anders Neijber, MD, Study Director — AstraZeneca
Locations (63):
- United States (63):
  - Research Site, Birmingham, Alabama
  - Research Site, Scottsdale, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Beverly Hills, California
  - Research Site, Burbank, California
  - Research Site, La Mesa, California
  - Research Site, Orange, California
  - Research Site, Pasadena, California
  - Research Site, San Diego, California
  - Research Site, Sherman Oaks, California
  - Research Site, Upland, California
  - Research Site, Wildomar, California
  - Research Site, New Britain, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Boca Raton, Florida
  - Research Site, Bradenton, Florida
  - Research Site, DeLand, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Fort Myers, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Maitland, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Tampa, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Edwardsville, Illinois
  - Research Site, Merrillville, Indiana
  - Research Site, Terre Haute, Indiana
  - Research Site, Newton, Kansas
  - Research Site, Prairie Village, Kansas
  - Research Site, Owensboro, Kentucky
  - Research Site, Lake Charles, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Haverhill, Massachusetts
  - Research Site, Okemos, Michigan
  - Research Site, Saint Paul, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Kenilworth, New Jersey
  - Research Site, Princeton, New Jersey
  - Research Site, Toms River, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, New York, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Toledo, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Eugene, Oregon
  - Research Site, Salem, Oregon
  - Research Site, Allentown, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Columbia, South Carolina
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Richmond, Virginia
  - Research Site, Kirkland, Washington
  - Research Site, Spokane, Washington
  - Research Site, Morgantown, West Virginia

REFERENCES:
- [Derived] Montgomery SA, Locklear JC, Svedsater H, Eriksson H. Efficacy of once-daily extended release quetiapine fumarate in patients with different levels of severity of generalized anxiety disorder. Int Clin Psychopharmacol. 2014 Sep;29(5):252-62. doi: 10.1097/YIC.0000000000000026. PMID 24394383
- [Derived] Stein DJ, Bandelow B, Merideth C, Olausson B, Szamosi J, Eriksson H. Efficacy and tolerability of extended release quetiapine fumarate (quetiapine XR) monotherapy in patients with generalised anxiety disorder: an analysis of pooled data from three 8-week placebo-controlled studies. Hum Psychopharmacol. 2011 Dec;26(8):614-28. doi: 10.1002/hup.1256. Epub 2011 Dec 6. PMID 22143997
- [Derived] Merideth C, Cutler AJ, She F, Eriksson H. Efficacy and tolerability of extended release quetiapine fumarate monotherapy in the acute treatment of generalized anxiety disorder: a randomized, placebo controlled and active-controlled study. Int Clin Psychopharmacol. 2012 Jan;27(1):40-54. doi: 10.1097/YIC.0b013e32834d9f49. PMID 22045039